CLINICAL TRIAL: NCT04209517
Title: Behavioral Markers of Pre-operative Anxiety : a Prospective Observational Study in Ambulatory Setting
Brief Title: Behavioral Markers of Pre-operative Anxiety
Acronym: KINESIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191092
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Preoperative Anxiety
Keywords: Preoperative anxiety; ethology; behavioural markers; objective detection
MeSH Terms: conditions — Behavior, Animal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Filming — Behavioural markers selection from video-recordings of the interview

SUMMARY:
The purpose of this study is to identify the characteristics of patients' behavioural patterns related to declared anxiety levels in a day-care surgical unit using ethological analysis of video-recordings of the pre-operative interview with the nurse.

DETAILED DESCRIPTION:
Guidelines in anaesthesia recommend systematic preoperative anxiety management to prevent negative perioperative impact, including impaired memory of important instructions and high incidence of post-operative acute and chronic pain. Self-administered questionnaires linked to scales to assess anxiety in the preoperative setting are usual practice. Yet, they are time consuming and rely on patient willingness to comply with instructions, which is not always reliable. The effects of acute anxiety on behaviour are poorly explored in the preoperative context. Quantifying and characterizing behavioural patterns in anxious patients using an applied ethological approach may provide useful information for reliable, accurate and objective assessment before surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for elective ambulatory surgery

Exclusion Criteria:

* communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective ambulatory surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between behaviour and anxiety | 1 day
  Correlation between behavioural markers and declarative anxiety

IPD SHARING:
Plan to Share IPD: No